CLINICAL TRIAL: NCT00511433
Title: A Randomized, Open-Label, Comparative Trial to Evaluate the Effects on Ovarian Function of a Monophasic Combined Oral Contraceptive (COC) Containing 2.5 mg Nomegestrol Acetate (NOMAC) and 1.5 mg Estradiol (E2), Compared to a Monophasic COC Containing 3 mg Drospirenone (DRSP) and 30 ug Ethinyl Estradiol (EE)
Brief Title: Effects on Ovarian Function of the Combined Oral Contraceptive NOMAC-E2 Compared to a COC Containing DRSP/EE (292003)(COMPLETED)(P05723)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P05723; Organon protocol 292003
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Results first posted 2011-08-29 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NOMAC-E2 (Experimental): Nomegestrol Acetate (NOMAC) and Estradiol (E2), 2.5 mg NOMAC and 1.5 mg E2 monophasic combined oral contraceptive
  Interventions: Drug: NOMAC-E2
- DRSP-EE (Active Comparator): Drospirenone (DRSP) and Ethinyl Estradiol (EE), 3 mg DRSP and 30 mcg EE monophasic combined oral contraceptive
  Interventions: Drug: DRSP-EE

INTERVENTIONS:
Drug: NOMAC-E2 — Nomegestrol Acetate and Estradiol Tablets, 2.5 mg NOMAC and 1.5 mg E2 taken once daily from Day 1 of menstrual period up to and including Day 28
  for 6 consecutive 28-day menstrual cycles.
  Arms: NOMAC-E2
Drug: DRSP-EE — Drospirenone and Ethinyl Estradiol Tablets, 3 mg DRSP and 30 mcg EE taken once daily from Day 1 of menstrual period up to and including Day 28 for 6 consecutive 28-day menstrual cycles.
  Arms: DRSP-EE

SUMMARY:
The primary purpose of this study is to evaluate the effects of the nomegestrol acetate-estradiol (NOMAC-E2) combined oral contraceptive (COC) on ovarian function.

ELIGIBILITY:
Inclusion Criteria:

* Willing to use COC for at least 6 cycles.
* 18 - 35 years of age at screening.
* Body Mass Index (BMI) of >/= 17 and </= 35.
* Good physical and mental health.
* Willing to use condoms as the sole contraceptive method during screening cycle and 1 post-treatment cycle.
* Willing to give informed consent.

Exclusion Criteria:

* Contraindications for contraceptive steroids (general).
* Additional contraindications (renal, hepatic or adrenal insufficiency).
* Breastfeeding.
* Present use (or use within 2 months prior to start of the trial medication) of the following drugs: phenytoin, barbiturates, primidone, carbamazepine, oxcarbazepine, topiramate, felbamate, rifampicin, nelfinavir, ritonavir, griseofulvin, ketoconazole, sex

steroids (other than pre- and post treatment contraceptive method) and herbal remedies containing Hypericum perforatum (St. John's Wort).

* Administration of any other investigational drugs and/or participation in another clinical trial within 2 months prior to the start of the trial medication or during the trial period.
* Abnormal cervical smear at screening, or documentation of an abnormal smear performed within 6 months before screening.
* Clinically relevant abnormal laboratory result at screening as judged by the investigator.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2006-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

REFERENCES:
- [Result] Duijkers IJ, Klipping C, Grob P, Korver T. Effects of a monophasic combined oral contraceptive containing nomegestrol acetate and 17 beta-oestradiol on ovarian function in comparison to a monophasic combined oral contraceptive containing drospirenone and ethinylestradiol. Eur J Contracept Reprod Health Care. 2010 Oct;15(5):314-25. doi: 10.3109/13625187.2010.504313. PMID 20695770

RESULTS

PARTICIPANT FLOW:
Groups:
- NOMAC-E2: Monophasic combined oral contraceptive (COC) tablets containing 2.5 mg Nomegestrol Acetate (NOMAC) and 1.5 mg Estradiol (E2) taken once daily from Day 1 of menstrual period up to and including Day 28 (Days 1-24, active tablets; Days 25-28, placebo tablets) for 6 consecutive 28-day menstrual cycles.
- DRSP-EE: Monophasic COC tablets containing 3 mg Drospirenone (DRSP) and 30 mcg Ethinyl Estradiol taken once daily from Day 1 of menstrual period up to and including Day 28 (Days 1-21, active tablets; Days 22-28, placebo tablets) for 6 consecutive 28-day menstrual cycles.
Period: Overall Study
Arm/Group | NOMAC-E2 | DRSP-EE
Started | 32 | 16
Completed | 26 | 15
Not Completed | 6 | 1
Not completed — Adverse Event | 5 | 0
Not completed — Other Reason | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NOMAC-E2 | DRSP-EE | Total
Number analyzed (Participants) | 32 | 16 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.8 (3.3) | 22.9 (4.3) | 22.8 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 16 | 48
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Effect on Cervical Mucus as Determined by Insler Score
Description: The Insler Score was assessed on Day 6 after ovulation during the Screening Cycle, on Day 21 of Cycle 1, and when the maximum follicle diameter was greater than or equal to 15 mm. The Insler Score consisted of four categories each scaled from 0 (none) to 3 (complete). The higher the score, the greater the cervical reaction.
Time Frame: Screening Cycle, Cycle 1, Cycle 2, and Cycle 7 (post-treatment cycle)
Population: ITT group consisted of all participants who were treated.
  n=number of participants with non-missing values at the respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 32 | 16
score on a scale
  Screening cycle (n=32 NOMAC-E2 / n=16 DRSP-EE) | 8.9 (2.55) | 7.3 (3.61)
  Cycle 1 (n=30 NOMAC-E2 / n=15 DRSP-EE) | 2.3 (1.93) | 3.2 (2.43)
  Cycle 2 (n=0 NOMAC-E2 / n=2 DRSP-EE) | NA (NA) — Mean and standard deviation do not apply for zero participants. | 4.5 (0.71)
  Cycle 7 (n=22 NOMAC-E2 / n=15 DRSP-EE) | 7.0 (2.94) | 8.7 (1.53)

2. Secondary Outcome: Effect on Maximum Endometrial Thickness
Description: Maximum endometrial thickness was defined as the largest endometrial thickness during a cycle.
Time Frame: Screening Cycle, Cycle 1, Cycle 2, and Cycle 6
Population: ITT group consisted of all participants who were treated.
  n=number of participants completing the respective cycle.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 32 | 16
mm
  Screening cycle (n=32 NOMAC-E2 / n=16 DRSP-EE) | 9.9 (1.91) | 10.1 (2.50)
  Cycle 1 (n=32 NOMAC-E2 / n=16 DRSP-EE) | 5.9 (1.22) | 6.1 (1.25)
  Cycle 2 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 5.3 (0.71) | 6.8 (1.73)
  Cycle 6 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 4.9 (0.66) | 5.5 (1.30)

3. Secondary Outcome: Number of In-treatment Pregnancies (With +2 Day Window) Per 100 Woman Years of Exposure (Pearl Index)
Description: In-treatment pregnancies were pregnancies with an estimated date of conception from the day of first intake of trial medication up to and including the day of last (active or placebo) intake of trial medication extended with a maximum of two days. Each 13 cycles (28 days per cycle) of exposure constitutes a woman year. The Pearl Index was obtained by dividing the number of in-treatment pregnancies that occurred by the time (in 100 woman years) that the women were under risk of becoming pregnant.
Time Frame: 6 cycles
Population: The "restricted ITT" set included all participants treated and excluded nonpregnant participants who didn't have >=1 cycle expected to be at risk for pregnancy (with recorded use of condoms or without sexual intercourse per diary card data).
Measure: Number (95% Confidence Interval); unit: Pregnancies per 100 woman years
Units Other Than Participants: woman years (rounded to nearest integer)
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 24 | 12
Number analyzed (woman years (rounded to nearest integer)) | 8 | 5
Pregnancies per 100 woman years | 0 [0 to 45.9] | 0 [0 to 72.7]

4. Secondary Outcome: Number of Participants With an Occurrence of Breakthrough Bleeding/Spotting
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary card booklets. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Breakthrough bleeding/spotting was defined as any episode that occurred during the "expected non-bleeding period" that was neither an early nor a continued withdrawal bleeding. Expected non-bleeding period: DRSP-EE group: 21-day period starting on Day 1 of the cycle; NOMAC-E2: 21-day period starting on Day 4 of the cycle.
Time Frame: Every 28-day cycle for 6 cycles
Population: The ITT group consisted of all participants who were treated; ITT analyses of vaginal bleeding patterns were based on all participants in the ITT group who had at least one evaluable cycle. Cycles were considered to be non-evaluable in case of insufficient bleeding data or improper cycle length.
  n=number of participants with evaluable cycles.
Measure: Number; unit: Participants
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 30 | 16
Participants
  Cycle 1 (n=30 NOMAC-E2 / n=16 DRSP-EE) | 7 | 1
  Cycle 2 (n=27 NOMAC-E2 / n=16 DRSP-EE) | 6 | 0
  Cycle 3 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 5 | 0
  Cycle 4 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 5 | 0
  Cycle 5 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 8 | 0
  Cycle 6 (n=26 NOMAC-E2 / n=14 DRSP-EE) | 5 | 0

5. Secondary Outcome: Number of Participants With an Occurrence of Absence of Withdrawal Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary card booklets. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Absence of withdrawal bleeding was defined as no bleeding/spotting episode that began during or continued into the "expected bleeding period". Expected bleeding period: DRSP-EE group: 7-day period starting on Day 22 of the cycle; NOMAC-E2: 7-day period starting on Day 25 of the cycle and ending on Day 3 of the next cycle.
Time Frame: Every 28-day cycle for 6 cycles
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 30 | 16
Participants
  Cycle 1 (n=30 NOMAC-E2 / n=16 DRSP-EE) | 3 | 0
  Cycle 2 (n=27 NOMAC-E2 / n=16 DRSP-EE) | 2 | 0
  Cycle 3 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 2 | 0
  Cycle 4 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 2 | 0
  Cycle 5 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 2 | 0
  Cycle 6 (n=26 NOMAC-E2 / n=14 DRSP-EE) | 4 | 1

6. Secondary Outcome: Number of Participants With an Occurrence of Breakthrough Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary card booklets. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Breakthrough bleeding was defined as any bleeding episode that occurred during the "expected non-bleeding period" that was neither part of an early nor continued withdrawal bleeding. Expected non-bleeding period: DRSP-EE group: 21-day period starting on Day 1 of the cycle; NOMAC-E2:21-day period starting on Day 4 of the cycle.
Time Frame: Every 28-day cycle for 6 cycles
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 30 | 16
Participants
  Cycle 1 (n=30 NOMAC-E2 / n=16 DRSP-EE) | 0 | 0
  Cycle 2 (n=27 NOMAC-E2 / n=16 DRSP-EE) | 0 | 0
  Cycle 3 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 0 | 0
  Cycle 4 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 1 | 0
  Cycle 5 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 1 | 0
  Cycle 6 (n=26 NOMAC-E2 / n=14 DRSP-EE) | 0 | 0

7. Secondary Outcome: Number of Participants With an Occurrence of Breakthrough Spotting (Spotting Only)
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary card booklets. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Breakthrough spotting was defined as any spotting episode that occurred during the "expected non-bleeding period" that was neither part of an early nor continued withdrawal bleeding. Expected non-bleeding period: DRSP-EE group: 21-day period starting on Day 1 of the cycle; NOMAC-E2:21-day period starting on Day 4 of the cycle.
Time Frame: Every 28-day cycle for 6 cycles
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 30 | 16
Participants
  Cycle 1 (n=30 NOMAC-E2 / n=16 DRSP-EE) | 7 | 1
  Cycle 2 (n=27 NOMAC-E2 / n=16 DRSP-EE) | 6 | 0
  Cycle 3 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 5 | 0
  Cycle 4 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 4 | 0
  Cycle 5 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 7 | 0
  Cycle 6 (n=26 NOMAC-E2 / n=14 DRSP-EE) | 5 | 0

8. Secondary Outcome: Number of Participants With an Occurrence of Early Withdrawal Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary card booklets. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Early withdrawal bleeding was defined as any withdrawal bleeding that started before the current "expected bleeding period". Expected bleeding period: DRSP-EE: 7-day period starting on Day 22 of the cycle; NOMAC-E2: 7-day period starting on Day 25 of the cycle and ending on Day 3 of the next cycle.
Time Frame: Every 28-day cycle for 6 cycles
Population: The ITT group consisted of all participants who were treated; ITT analyses of vaginal bleeding patterns were based on all participants in the ITT group who had at least one evaluable cycle. Cycles were considered to be non-evaluable in case of insufficient bleeding data or improper cycle length.
  n= number of participants with evaluable cycles.
Measure: Number; unit: Participants
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 30 | 16
Participants
  Cycle 1 (n=30 NOMAC-E2 / n=16 DRSP-EE) | 4 | 2
  Cycle 2 (n=27 NOMAC-E2 / n=16 DRSP-EE) | 4 | 0
  Cycle 3 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 1 | 0
  Cycle 4 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 2 | 0
  Cycle 5 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 1 | 0
  Cycle 6 (n=26 NOMAC-E2 / n=14 DRSP-EE) | 2 | 0

9. Secondary Outcome: Number of Participants With an Occurrence of Continued Withdrawal Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary card booklets. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Continued withdrawal bleeding was defined as any withdrawal bleeding that continued into the "expected non-bleeding period" of the next cycle. Expected non-bleeding period: DRSP-EE group: 21-day period starting on Day 1 of the cycle; NOMAC-E2: 21-day period starting on Day 4 of the cycle.
Time Frame: Every 28-day cycle for 5 cycles
Population: The ITT group consisted of all participants who were treated; ITT analyses of vaginal bleeding patterns were based on all participants in the ITT group who had at least one evaluable cycle. Cycles were considered to be non-evaluable in case of insufficient bleeding data or improper cycle length.
Measure: Number; unit: Participants
Groups:
- NOMAC-E2: Monophasic combined oral contraceptive (COC) tablets containing 2.5 mg Nomegestrol Acetate (NOMAC) and 1.5 mg Estradiol (E2) taken once daily from Day 1 of menstrual period up to and including Day 28 (Days 1-24, active tablets; Days 25-28, placebo tablets) for 6 consecutive 28-day menstrual cycles.
  n=number of participants with evaluable cycles (except for the very last cycle of a participant for which this parameter was not defined).
- DRSP-EE: Monophasic COC tablets containing 3 mg Drospirenone (DRSP) and 30 mcg Ethinyl Estradiol taken once daily from Day 1 of menstrual period up to and including Day 28 (Days 1-21, active tablets; Days 22-28, placebo tablets) for 6 consecutive 28-day menstrual cycles.
  n=number of participants with evaluable cycles (except for the very last cycle of a participant for which this parameter was not defined).
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 30 | 16
Participants
  Cycle 1 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 11 | 12
  Cycle 2 (n=27 NOMAC-E2 / n=16 DRSP-EE) | 8 | 10
  Cycle 3 (n=25 NOMAC-E2 / n=15 DRSP-EE) | 8 | 11
  Cycle 4 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 12 | 12
  Cycle 5 (n=26 NOMAC-E2 / n=14 DRSP-EE) | 9 | 10

10. Primary Outcome: Effect on Ovarian Function as Determined by the Number of Participants With an Occurrence of Ovulation
Description: During treatment, ovulation was assessed for each participant by the investigator on the basis of ultrasound scanning (USS). The final analysis was based on assessor-blind adjudication.
Time Frame: Cycle 1, Cycle 2, and Cycle 6
Population: Intent-to-treat (ITT) group consisted of all participants who were treated.
  n=number of participants completing the respective cycle with non-missing values.
Measure: Number; unit: Participants
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 32 | 16
Participants
  Cycle 1 (n=32 NOMAC-E2 / n=16 DRSP-EE) | 0 | 0
  Cycle 2 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 0 | 0
  Cycle 6 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 0 | 0

11. Primary Outcome: Effect on Ovarian Function as Determined by the Maximum Follicle Diameter
Description: The maximum follicular diameter was defined as the largest follicular diameter during a treatment cycle.
Time Frame: Screening cycle, Cycle 1, Cycle 2, Cycle 3, and Cycle 6
Population: ITT group consisted of all participants who were treated.
  n=number of participants completing the respective cycle with non-missing values.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 32 | 16
millimeters (mm)
  Screening cycle (n=32 NOMAC-E2 / n=16 DRSP-EE) | 19.3 (3.13) | 19.6 (4.32)
  Cycle 1 (n=32 NOMAC-E2 / n=16 DRSP-EE) | 7.6 (1.51) | 8.1 (1.98)
  Cycle 2 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 8.2 (1.82) | 10.8 (4.76)
  Cycle 3 (n=27 NOMAC-E2 / n=14 DRSP-EE) | 7.8 (1.88) | 8.4 (2.31)
  Cycle 6 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 6.9 (2.07) | 7.4 (2.06)

12. Primary Outcome: Effect on Ovarian Function as Determined by the Maximum Progesterone Value
Description: The maximum progesterone value was defined as the largest value during a cycle.
Time Frame: Screening cycle, Cycle 1, Cycle 2, Cycle 3, and Cycle 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 32 | 16
nanomoles per liter (nmol/L)
  Screening cycle (n=32 NOMAC-E2 / n=16 DRSP-EE) | 38.7 (12.62) | 38.7 (17.01)
  Cycle 1 (n=32 NOMAC-E2 / n=16 DRSP-EE) | 1.7 (0.46) | 1.6 (0.28)
  Cycle 2 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 1.5 (0.46) | 1.5 (0.26)
  Cycle 3 (n=27 NOMAC-E2 / n=14 DRSP-EE) | 1.26 (0.10) | 1.34 (0.27)
  Cycle 6 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 1.3 (0.29) | 1.5 (0.26)

13. Primary Outcome: Effect on Ovarian Function as Determined by 17 Beta-estradiol (E2)
Description: The parameter was measured at pre-defined study days.
Time Frame: Cycle 1, Cycle 2, Cycle 3, and Cycle 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: picomoles per liter (pmol/L)
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 32 | 16
picomoles per liter (pmol/L)
  Cycle 1, Day 2 (n=32 NOMAC-E2 / n=16 DRSP-EE) | 168.75 (62.37) | 79.82 (18.34)
  Cycle 1, Day 5 (n=32 NOMAC-E2 / n=16 DRSP-EE) | 194.57 (93.17) | 66.66 (10.53)
  Cycle 1, Day 8 (n=32 NOMAC-E2 / n=16 DRSP-EE) | 172.35 (66.92) | 61.15 (3.66)
  Cycle 1, Day 11 (n=30 NOMAC-E2 / n=16 DRSP-EE) | 184.63 (95.70) | 60.51 (1.96)
  Cycle 1, Day 14 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 197.57 (123.23) | 60.26 (1.48)
  Cycle 1, Day 18 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 182.72 (84.03) | 60.58 (2.93)
  Cycle 1, Day 21 (n=30 NOMAC-E2 / n=16 DRSP-EE) | 191.08 (139.50) | 59.82 (0)
  Cycle 1, Day 24 (n=30 NOMAC-E2 / n=16 DRSP-EE) | 232.80 (281.15) | 69.84 (23.50)
  Cycle 1, Day 27 (n=30 NOMAC-E2 / n=16 DRSP-EE) | 99.65 (42.53) | 150.79 (46.45)
  Cycle 2, Day 2 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 176.43 (91.99) | 135.86 (106.62)
  Cycle 2, Day 5 (n=29 NOMAC-E2 / n=15 DRSP-EE) | 213.64 (104.85) | 142.74 (186.99)
  Cycle 2, Day 8 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 192.59 (68.83) | 131.98 (196.51)
  Cycle 2, Day 11 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 185.77 (63.97) | 112.23 (152.19)
  Cycle 2, Day 14 (n=29 NOMAC-E2 / n=15 DRSP-EE) | 183.66 (74.39) | 78.44 (69.99)
  Cycle 2, Day 18 (n=28 NOMAC-E2 / n=15 DRSP-EE) | 213.84 (123.35) | 60.11 (0.95)
  Cycle 2, Day 21 (n=27 NOMAC-E2 / n=16 DRSP-EE) | 192.47 (66.43) | 59.91 (0.37)
  Cycle 2, Day 24 (n=27 NOMAC-E2 / n=16 DRSP-EE) | 206.20 (147.27) | 61.33 (3.95)
  Cycle 2, Day 27 (n=27 NOMAC-E2 / n=16 DRSP-EE) | 97.99 (40.88) | 155.63 (63.65)
  Cycle 3, Day 2 (n=27 NOMAC-E2 / n=14 DRSP-EE) | 148.16 (52.09) | 141.11 (115.89)
  Cycle 6, Day 14 (n=25 NOMAC-E2 / n=14 DRSP-EE) | 205.89 (104.45) | 59.98 (0.59)
  Cycle 6, Day 18 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 200.04 (90.28) | 64.20 (12.99)
  Cycle 6, Day 21 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 188.47 (90.12) | 60.82 (3.02)
  Cycle 6, Day 24 (n=26 NOMAC-E2 / n=14 DRSP-EE) | 187.16 (106.60) | 69.60 (33.97)
  Cycle 6, Day 27 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 99.51 (35.60) | 133.49 (61.28)

14. Primary Outcome: Effect on Ovarian Function as Determined by Follicle Stimulating Hormone (FSH)
Description: The parameter was measured at pre-defined study days.
Time Frame: Cycle 1, Cycle 2, Cycle 3, and Cycle 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 32 | 16
International units per liter (IU/L)
  Cycle 1, Day 2 (n=32 NOMAC-E2 / n=16 DRSP-EE) | 4.29 (1.45) | 4.51 (1.14)
  Cycle 1, Day 5 (n=32 NOMAC-E2 / n=16 DRSP-EE) | 4.08 (1.59) | 4.23 (1.33)
  Cycle 1, Day 8 (n=32 NOMAC-E2 / n=16 DRSP-EE) | 3.59 (1.59) | 3.40 (1.57)
  Cycle 1, Day 11 (n=30 NOMAC-E2 / n=16 DRSP-EE) | 3.44 (2.07) | 2.46 (1.40)
  Cycle 1, Day 14 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 3.06 (1.90) | 2.32 (1.71)
  Cycle 1, Day 18 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 2.95 (1.76) | 1.91 (1.69)
  Cycle 1, Day 21 (n=30 NOMAC-E2 / n=16 DRSP-EE) | 2.87 (1.96) | 1.61 (1.53)
  Cycle 1, Day 24 (n=30 NOMAC-E2 / n=16 DRSP-EE) | 2.88 (1.99) | 4.50 (4.05)
  Cycle 1, Day 27 (n=30 NOMAC-E2 / n=16 DRSP-EE) | 5.42 (2.51) | 7.91 (3.95)
  Cycle 2, Day 2 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 5.32 (2.05) | 5.48 (1.82)
  Cycle 2, Day 5 (n=29 NOMAC-E2 / n=15 DRSP-EE) | 4.59 (1.54) | 4.08 (1.54)
  Cycle 2, Day 8 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 3.99 (1.71) | 2.77 (1.19)
  Cycle 2, Day 11 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 3.47 (1.68) | 1.96 (1.13)
  Cycle 2, Day 14 (n=29 NOMAC-E2 / n=15 DRSP-EE) | 3.34 (2.18) | 1.44 (1.00)
  Cycle 2, Day 18 (n=28 NOMAC-E2 / n=15 DRSP-EE) | 3.18 (1.84) | 1.22 (0.94)
  Cycle 2, Day 21 (n=27 NOMAC-E2 / n=16 DRSP-EE) | 3.02 (1.64) | 1.04 (0.98)
  Cycle 2, Day 24 (n=27 NOMAC-E2 / n=16 DRSP-EE) | 3.05 (1.76) | 3.52 (3.51)
  Cycle 2, Day 27 (n=27 NOMAC-E2 / n=16 DRSP-EE) | 5.92 (2.77) | 6.99 (2.78)
  Cycle 3, Day 2 (n=27 NOMAC-E2 / n=14 DRSP-EE) | 6.01 (2.08) | 5.17 (1.44)
  Cycle 6, Day 14 (n=25 NOMAC-E2 / n=14 DRSP-EE) | 3.08 (1.88) | 1.43 (1.32)
  Cycle 6, Day 18 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 2.82 (1.79) | 1.29 (1.28)
  Cycle 6, Day 21 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 3.30 (2.14) | 0.92 (0.96)
  Cycle 6, Day 24 (n=26 NOMAC-E2 / n=14 DRSP-EE) | 2.86 (2.09) | 3.18 (3.04)
  Cycle 6, Day 27 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 5.65 (2.57) | 6.22 (2.99)

15. Secondary Outcome: Average Number of Breakthrough Bleeding/Spotting Days
Description: as for outcome 4
Time Frame: Every 28-day cycle for 6 cycles
Population: ITT analyses of vaginal bleeding patterns were based on all participants in the ITT group who had at least one evaluable cycle. Cycles were considered to be non-evaluable in case of insufficient bleeding data or improper cycle length.
  n= number of participants who had breakthrough bleeding/spotting for the respective cycle.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 30 | 16
Days
  Cycle 1 (n=7 NOMAC-E2; n=1 DRSP-EE) | 3.0 (2.2) | 2.0 (NA) — Value for one participant; therefore, standard deviation does not apply.
  Cycle 2 (n=6 NOMAC-E2; n=0 DRSP-EE) | 2.7 (1.9) | NA (NA) — Mean and standard deviation do not apply for zero participants.
  Cycle 3 (n=5 NOMAC-E2; n=0 DRSP-EE) | 2.2 (1.1) | NA (NA) — Mean and standard deviation do not apply for zero participants.
  Cycle 4 (n=5 NOMAC-E2; n=0 DRSP-EE) | 4.0 (2.8) | NA (NA) — Mean and standard deviation do not apply for zero participants.
  Cycle 5 (n=8 NOMAC-E2; n=0 DRSP-EE) | 3.5 (2.3) | NA (NA) — Mean and standard deviation do not apply for zero participants.
  Cycle 6 (n=5 NOMAC-E2; n=0 DRSP-EE) | 3.6 (2.1) | NA (NA) — Mean and standard deviation do not apply for zero participants.

16. Secondary Outcome: Average Number of Withdrawal Bleeding Days
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using diary card booklets. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Withdrawal bleeding was defined as bleeding/spotting episode that started during or continued into the "expected bleeding period". Expected bleeding period: DRSP-EE group: 7-day period starting on Day 22 of the cycle; NOMAC-E2: 7-day period starting on Day 25 of the cycle and ending on Day 3 of the next cycle.
Time Frame: Every 28-day cycle for 6 cycles
Population: ITT analyses of vaginal bleeding patterns were based on all participants in the ITT group who had at least one evaluable cycle. Cycles were considered to be non-evaluable in case of insufficient bleeding data or improper cycle length.
  n= number of participants who had withdrawal bleeding/spotting for the respective cycle.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 30 | 16
Days
  Cycle 1 (n=27 NOMAC-E2; n=16 DRSP-EE) | 7.2 (6.7) | 7.0 (4.7)
  Cycle 1 (n=25 NOMAC-E2; n=16 DRSP-EE) | 7.4 (7.5) | 5.0 (1.7)
  Cycle 3 (n=24 NOMAC-E2; n=15 DRSP-EE) | 4.3 (2.4) | 5.4 (1.5)
  Cycle 4 (n=24 NOMAC-E2; n=15 DRSP-EE) | 4.7 (1.9) | 5.3 (1.0)
  Cycle 5 (n=24 NOMAC-E2; n=15 DRSP-EE) | 5.5 (6.1) | 4.9 (1.1)
  Cycle 6 (n=22 NOMAC-E2; n=13 DRSP-EE) | 5.2 (6.3) | 3.9 (0.9)

17. Primary Outcome: Effect on Ovarian Function as Determined by Luteinizing Hormone (LH)
Description: The parameter was measured at pre-defined study days.
Time Frame: Cycle 1, Cycle 2, Cycle 3, and Cycle 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 32 | 16
IU/L
  Cycle 1, Day 2 (n=32 NOMAC-E2 / n=16 DRSP-EE) | 3.73 (1.64) | 3.69 (1.58)
  Cycle 1, Day 5 (n=32 NOMAC-E2 / n=16 DRSP-EE) | 2.98 (1.49) | 4.34 (2.35)
  Cycle 1, Day 8 (n=32 NOMAC-E2 / n=16 DRSP-EE) | 2.50 (1.68) | 3.09 (2.36)
  Cycle 1, Day 11 (n=30 NOMAC-E2 / n=16 DRSP-EE) | 2.13 (1.50) | 1.89 (1.45)
  Cycle 1, Day 14 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 1.85 (1.77) | 2.32 (2.05)
  Cycle 1, Day 18 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 1.76 (1.41) | 1.61 (1.29)
  Cycle 1, Day 21 (n=30 NOMAC-E2 / n=16 DRSP-EE) | 1.45 (1.33) | 1.19 (0.86)
  Cycle 1, Day 24 (n=30 NOMAC-E2 / n=16 DRSP-EE) | 1.59 (1.44) | 2.63 (2.07)
  Cycle 1, Day 27 (n=30 NOMAC-E2 / n=16 DRSP-EE) | 3.04 (1.95) | 4.34 (2.38)
  Cycle 2, Day 2 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 3.47 (2.20) | 4.81 (3.01)
  Cycle 2, Day 5 (n=29 NOMAC-E2 / n=15 DRSP-EE) | 3.04 (1.94) | 5.08 (3.21)
  Cycle 2, Day 8 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 2.48 (1.85) | 3.33 (1.97)
  Cycle 2, Day 11 (n=29 NOMAC-E2 / n=16 DRSP-EE) | 2.54 (2.01) | 2.70 (2.18)
  Cycle 2, Day 14 (n=29 NOMAC-E2 / n=15 DRSP-EE) | 2.39 (2.17) | 1.69 (1.42)
  Cycle 2, Day 18 (n=28 NOMAC-E2 / n=15 DRSP-EE) | 2.05 (1.76) | 1.60 (1.31)
  Cycle 2, Day 21 (n=27 NOMAC-E2 / n=16 DRSP-EE) | 1.68 (1.44) | 0.97 (0.67)
  Cycle 2, Day 24 (n=27 NOMAC-E2 / n=16 DRSP-EE) | 1.81 (1.75) | 2.38 (2.01)
  Cycle 2, Day 27 (n=27 NOMAC-E2 / n=16 DRSP-EE) | 3.37 (2.90) | 3.92 (2.17)
  Cycle 3, Day 2 (n=27 NOMAC-E2 / n=14 DRSP-EE) | 3.71 (2.23) | 4.79 (2.67)
  Cycle 6, Day 14 (n=25 NOMAC-E2 / n=14 DRSP-EE) | 2.29 (1.86) | 2.15 (2.83)
  Cycle 6, Day 18 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 1.88 (2.05) | 1.27 (1.02)
  Cycle 6, Day 21 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 2.00 (1.68) | 1.14 (0.89)
  Cycle 6, Day 24 (n=26 NOMAC-E2 / n=14 DRSP-EE) | 1.85 (1.75) | 2.56 (2.12)
  Cycle 6, Day 27 (n=26 NOMAC-E2 / n=15 DRSP-EE) | 3.13 (2.21) | 4.03 (2.57)

ADVERSE EVENTS:
Arm/Group | NOMAC-E2 | DRSP-EE
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/16
Other Adverse Events (participants affected / at risk) | 30/32 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOMAC-E2 (N=32) | DRSP-EE (N=16)
Appendicitis perforated (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOMAC-E2 (N=32) | DRSP-EE (N=16)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 5 (6) | 3 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 11 (13) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (11) | 3 (5)
Toothache (Gastrointestinal disorders) | 3 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (5)
Fatigue (General disorders) | 2 (2) | 1 (1)
Hangover (General disorders) | 5 (7) | 1 (1)
Malaise (General disorders) | 3 (3) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 4 (8) | 3 (4)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 5 (7) | 7 (7)
Nasopharyngitis (Infections and infestations) | 15 (23) | 9 (12)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Vaginal candidiasis (Infections and infestations) | 2 (2) | 1 (1)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 0 (0)
Weight increased (Investigations) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (8) | 1 (2)
Dizziness (Nervous system disorders) | 3 (4) | 0 (0)
Headache (Nervous system disorders) | 8 (17) | 4 (7)
Affect lability (Psychiatric disorders) | 4 (4) | 1 (1)
Depressed mood (Psychiatric disorders) | 3 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 1 (1)
Breast enlargement (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 4 (7)
Breast tenderness (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 3 (4) | 2 (2)
Vaginal discharge (Reproductive system and breast disorders) | 2 (2) | 1 (3)
Vaginal odour (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor recognizes the right of the investigator(s) to publish, but all publications must be based on data validated and released by the Sponsor. Any such scientific paper, presentation, or other communication concerning the clinical trial will first be submitted to the Sponsor, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.